CLINICAL TRIAL: NCT02994407
Title: Safety, Tolerability, and Pharmacokinetics Study of Single and Multiple Subcutaneous Doses of Turoctocog Alfa Pegol in Patients With Haemophilia A
Brief Title: Safety, Tolerability, and Pharmacokinetics Study of Turoctocog Alfa Pegol Injected Under the Skin in Patients With Haemophilia A
Acronym: alleviate 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7170-4213; U1111-1183-5111 (Other: WHO); 2016-002396-99 (EudraCT Number); JapicCTI-173683 (Registry Identifier: JAPIC)
Record Dates: First submitted 2016-12-13; First posted 2016-12-15 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- N8-GP s.c. (Experimental)
  Interventions: Drug: turoctocog alfa pegol

INTERVENTIONS:
Drug: turoctocog alfa pegol — Part A: Participants will receive a single dose of turoctocog alfa pegol, administered subcutaneously (under the skin), at a dose of 12.5, 25 or 50 U/kg.
  Part B: Participants will receive a daily dose of turoctocog alfa pegol, as identified in Part A, as a subcutaneous (under the skin) injection for a period of 3 months.

SUMMARY:
The trial is conducted in Asia, Europe and North America. The aim of the study is to evaluate the safety of administration under the skin of turoctocog alfa pegol (SC N8-GP) in patients with severe haemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Male, age above or equal to 18 years at the time of signing informed consent,(part A).
* Male, age above or equal to 12 years at the time of signing informed consent,(part B).
* Diagnosis of congenital haemophilia A based on medical records (FVIII activity <1%).
* History of more than 150 exposure days to any FVIII containing products.

Exclusion Criteria:

* Previous participation in this trial. Participation is defined as signed informed consent.

(Patients who have completed part A are allowed to also participate in part B. If so, a separate informed consent covering part B must be signed.)

* Immune compromised patients due to human immunodeficiency virus (HIV) infection (defined as viral load greater than or equal to 400.000 copies/mL and/or cluster of differentiation 4+ (CD4+) lymphocyte count less than or equal to 200/μL performed at screening or defined by medical records no older than 6 months)
* Any history of FVIII inhibitors (defined by medical records within 8 years of randomisation)
* Inhibitors to FVIII (greater than or equal to 0.6 Bethesda unit (BU)) at screening, measured by Nijmegen modified Bethesda method at central laboratory.

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | Day 0-Day 28
  Count and % of Adverse events

SECONDARY OUTCOMES:
Cmax | 0-144 hours
  Calculated based on plasma FVIII activity measured in blood.
Incidence of FVIII inhibitors above or equal to 0.6 BU | Day 0-Day 28
  Count of presence of inhibitors
Area under the activity time curve from 0 to infinity | 0-144 hours
  Calculated based on plasma FVIII activity measured in blood.
Area under the activity time curve from 0 to t | 0-144 hours
  Calculated based on plasma FVIII activity measured in blood.
Area under the activity time curve from 0 to last | 0-144 hours
  Calculated based on plasma FVIII activity measured in blood.
tmax- time to maximal FVIII activity | 0-144 hours
  Calculated based on plasma FVIII activity measured in blood.
Cmin -the minimal FVIII activity | 0-144 hours
  Calculated based on plasma FVIII activity measured in blood.
tmin - time to minimal FVIII activity | 0-144 hours
  Calculated based on plasma FVIII activity measured in blood.
Css, min - the minimum FVIII activity at steady state | 0-144 hours
  Calculated based on plasma FVIII activity measured in blood.
Css, max - the maximal FVIII activity at steady state | 0-144 hours
  Calculated based on plasma FVIII activity measured in blood.
Css - the mean FVIII activity at steady state | 0-144 hours
  Calculated based on plasma FVIII activity measured in blood.
Racc - accumulation ratio | 0-144 hours
  Calculated based on plasma FVIII activity measured in blood.
t½ - terminal half-life | 0-144 hours
  Calculated based on plasma FVIII activity measured in blood.
CL - total plasma clearance of drug after intravenous administration | 0-144 hours
  Calculated based on plasma FVIII activity measured in blood.
Vz -apparent volume of distribution during terminal phase | 0-144 hours
  Calculated based on plasma FVIII activity measured in blood.
Vss - apparent volume of distribution during steady state | 0-144 hours
  Calculated based on plasma FVIII activity measured in blood.
MRT - mean residence time | 0-144 hours
  Calculated based on plasma FVIII activity measured in blood.
Injection site reactions | Day 0 - day 28
  Count of reactions
Number of treatment requiring bleeding episodes | Day 0 - day 120
  Count of episodes
Consumption of FVIII | Day 0 - day 120
  Measured in IU
Change in Coagulation parameters, fibrinogen | Day 0, day 7
  Measured in g/L
Change in Coagulation parameters, antithrombin | Day 0, day 7
  Measured in %
Change in Coagulation parameters, international normalised ratio | Day 0, day 7
  Measured in INR
Change in Coagulation parameters, activated partial thromboplastin time | Day 0, day 7
  Measured in sec.
Change in Coagulation parameters, von Willebrand Factor | Day 0, day 7
  Measured in %

CONTACTS AND LOCATIONS:
Locations (18):
- United States (8):
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, East Lansing, Michigan
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Norfolk, Virginia
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Austria (2):
  - Novo Nordisk Investigational Site, Innsbruck
  - Novo Nordisk Investigational Site, Vienna
- Novo Nordisk Investigational Site, Nantes, France
- Germany (3):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Duisburg
  - Novo Nordisk Investigational Site, Homburg
- Japan (2):
  - Novo Nordisk Investigational Site, Shinjuku-ku, Tokyo
  - Novo Nordisk Investigational Site, Tokyo
- Serbia (2):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Novi Sad

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Derived] Klamroth R, Feistritzer C, Friedrich U, Lentz SR, Reichwald K, Zak M, Chowdary P. Pharmacokinetics, immunogenicity, safety, and preliminary efficacy of subcutaneous turoctocog alfa pegol in previously treated patients with severe hemophilia A (alleviate 1). J Thromb Haemost. 2020 Feb;18(2):341-351. doi: 10.1111/jth.14660. Epub 2019 Nov 15. PMID 31618804